CLINICAL TRIAL: NCT02474004
Title: 3D-gait Analysis in Patients With Medial Meniscus Repair vs. Partial Meniscectomy
Brief Title: Gait Analysis Meniscal Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Michael Liebensteiner (Other)
Responsible Party: Sponsor-Investigator, Michael Liebensteiner, Physician, Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: GAIT-Men1
Record Dates: First submitted 2015-06-04; First posted 2015-06-17 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Lesion of the Medial Meniscus

ARMS (2):
- medial meniscus repair (Experimental): patients receiving medial meniscus repair
  Interventions: Procedure: medial meniscal surgery
- medial partial meniscectomy (Active Comparator): patients having medial partial meniscectomy
  Interventions: Procedure: medial meniscal surgery

INTERVENTIONS:
Procedure: medial meniscal surgery — one group/arm has meniscal repair as part of clinical routine one group/arm has meniscal partial resection as part of clinical routine both groups have gait analysis & knee scores 6 mo after the procedures

SUMMARY:
In the past it was shown, that medial partial meniscectomy (MPM) leads to an increase of the knee adduction moment (KAM) during walking. Other researches found out that an increase of the KAM is an important factor contributing to degeneration joint disease of the knee (osteoarthritis). Today, medial menicus repair (MMR) is favoured by many knee surgeons, because preserving as much of the meniscus as possible is assumed to delay degenerative joint disease.

The investigators hypothesize significant differences in knee adduction moments between patients treated with partial medial meniscectomy vs. patients treated with medial meniscus repair (hypothesis 1; major hypothesis). Additionally, it is hypothesized that: the mentioned groups differ with respect to other kinetic and kinematic key parameters of gait (hypothesis 2) and that the knee adduction moment correlates with the clinical outcome as determined by a typical knee score (hypothesis 3).

ELIGIBILITY:
Inclusion Criteria: patients with traumatic medial meniscus lesions scheduled for meniscal repair or resection

Exclusion Criteria:

* previous or current diseases of the back and the other joints of the lower limbs
* any form of inflammatory arthritis
* diabetes
* neurological disorders
* other conditions that may affect gait

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-02; Primary Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
knee adduction moment [Nm/kg] | once after 6 months
  a parameter of gait analysis

SECONDARY OUTCOMES:
set of kinetic, kinematic and temporospatial gait parameters | once after 6 months
  other gait parameters

OTHER OUTCOMES:
KOOS | 6 months post
  knee specific patient-reported outcome measurement

CONTACTS AND LOCATIONS:
Locations (2):
- Austria (2):
  - Innsbruck Medical University, Dept. Orthop. Surgery, Innsbruck, Tyrol
  - Sportsclinic Austria, Innsbruck, Tyrol